CLINICAL TRIAL: NCT06334510
Title: Phase IV Clinical Study on Safety and Efficacy of Quadrivalent Influenza Virus Split Vaccine in Larger Population
Brief Title: Evaluate the Safety and Efficacy of Quadrivalent Influenza in Real-world Situations.
Status: Completed | Type: Observational
Sponsor: Hualan Biological Bacterin Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-SJLG-2021-Ⅳ-01
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: GCP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 3ml of blood was collected before and 30 days after immunization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Approval consistency study: A total of 1050 recipients aged 18-59 years were enrolled in this study. Blood samples were collected before and 30 days after vaccination. Hemagglutination inhibition (HI) antibody to influenza virus was detected in the serum of all recipients to evaluate the inter-batch consistency of the vaccine.
  Interventions: Biological: One dose of quadrivalent influenza virus split vaccine was administered
- Safety and immunogenicity in a larger vaccination cohort aged 3 years and older: 3850 recipients were enrolled in an open trial: safety observation after vaccination, follow-up for adverse events (AE) 30 minutes and 0-30 days after vaccination, and SAEs for 6 months after vaccination.
  Interventions: Biological: One dose of quadrivalent influenza virus split vaccine was administered

INTERVENTIONS:
Biological: One dose of quadrivalent influenza virus split vaccine was administered — Safety observation: All 4900 vaccine recipients participated in the safety observation after vaccination, and were followed up for adverse events (AE) within 30 minutes and 0-30 days after vaccination, and SAEs within 6 months after vaccination.
  In addition to 1050 recipients aged 18-59 years who were included in the first layer test, 350 recipients aged 3-17 years and 350 recipients aged ≥60 years were randomly selected from each group. Blood samples were collected before and 30 days after vaccination for influenza virus HI antibody detection.

SUMMARY:
To evaluate the inter-batch consistency (CI) of quadrivalent influenza vaccine (split virion) among healthy people aged 18-59 years； Secondly, to evaluate the safety and immunogenicity of quadrivalent influenza vaccine (split virion) in the expanded population aged 3 years and above, in order to observe the rare adverse reaction of 1‰.

DETAILED DESCRIPTION:
The study was divided into two parts. The first part was an inter-batch consistency study (a randomized, double-blind, 1050 subjects aged 18-59 years). The second part was the safety and immunogenicity study in the expanded population aged 3 years and above (enrollment 4900).were selected to receive of normal commercially available quadrivalent influenza vaccine。 Safety observation: follow-up was conducted to observe the occurrence of AE within 30 minutes (0 day) and 0-30 days after vaccination, and the occurrence of SAE within 6 months after vaccination.

Immunogenicity observation: Blood samples were collected from all subjects before and 30 days after vaccination for influenza virus HI antibody detection。 According to the European Union seasonal influenza evaluation criteria, if the HI antibody seroconversion rate of each subtype of influenza virus was ≥40%, the HI antibody positive rate was ≥70%, and the GMI of each subtype of influenza virus was ≥2.5 times 30 days after any dose of vaccination, the vaccination schedule was considered to have acceptable immunogenicity.

Safety outcome MEASURES The occurrence of adverse reactions/events after each dose of vaccination was observed. The incidence of ① total adverse reactions/events, ② incidence of grade 3 or above adverse reactions/events and SAE, ③ incidence of adverse reactions/events severity classification, ④ incidence of adverse reactions/events by type (inoculation site and systemic, SOC, PT) and incidence of adverse reactions/events severity classification were calculated.

Note: Known adverse effects of quadrivalent influenza vaccine that have been identified in previous clinical studies are as follows:

Inoculation site (local) adverse events: pain, induration, swelling, rash, redness, pruritus, cellulitis.

Adverse events at non-inoculated sites (systemic) included fever, diarrhea, constipation, dysphagia, anorexia, vomiting, nausea, myalgia (non-inoculated sites), arthralgia, headache, cough, dyspnea, pruritus at non-inoculated sites (without skin lesions), mucocutaneous abnormalities, irritation/inhibition, acute anaphylaxis, and fatigue/fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people aged 3 years and above;
* I (or/and his/her legal guardian/authorized representative) can comply with the requirements of the clinical trial protocol after informed consent and voluntary signed informed consent;
* No contraindications of quadrivalent influenza vaccine in the package insert and meet the vaccination requirements after medical history inquiry.

Exclusion Criteria:

* Allergy to any component of the quadrivalent influenza vaccine, including egg, excipients, formaldehyde, or Triton X-100;
* people with a history of anaphylaxis after vaccination (allergy to any previous vaccination);
* Acute disease, severe chronic disease, acute onset of chronic disease, cold and fever;
* Axillary body temperature ≥37.3℃ (> 14 years old) and ≥37.5℃ (≤14 years old) before vaccination;
* Uncontrolled epilepsy;
* patients with progressive neurological disease or a history of Guillain-Barre syndrome;
* receiving immunoglobulin injection for less than one month;
* vaccination with live attenuated vaccine within 14 days before and other vaccines within 7 days before vaccination;

Ages: 3 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy people aged 3 years and older
Sampling Method: Probability Sample
Enrollment: 4900 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and immunogenicity of Hualan Biovar quadrivalent influenza vaccine in a larger population in the real world, and to observe rare adverse drug reaction (ADR) of 1‰. | The safety was observed until 6 months after the full course of immunization
  The incidence of adverse events/reactions after quadrivalent influenza vaccination was observed, and the incidence of ① total adverse events/reactions, ② incidence of grade 3 or above adverse events/reactions and SAE, ③ incidence of adverse events/reactions according to severity classification of adverse events/reactions and ④ incidence of symptomatic adverse events/reactions were calculated.

SECONDARY OUTCOMES:
To explore the consistency of three consecutive batches of commercial vaccines for vaccination in adults aged 18-59 years. | Before and 30 days after immunization
  The lower limit of the 95% confidence interval (CI) of the seroconversion rate (SCR) of hemagglutination inhibition (HAI) antibodies against each virus strain after vaccination was ≥40%. The lowest dilution used in the assay was 1 in 10. Seroconversion was defined as a prevaccination HAI titer of <1:10 and a postvaccination titer of ≥1:40 or a prevaccination titer of ≥1:10 and a 4-fold or greater increase in titer after vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Kou Zengqiang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided